CLINICAL TRIAL: NCT06047548
Title: A Phase 3b, Randomized Controlled Study to Evaluate the Efficacy and Safety of Tirzepatide Once Weekly 5 mg and/or Maximum Tolerated Dose Versus Placebo for Maintenance of Body Weight Reduction in Participants Who Have Obesity or Overweight With Weight-Related Comorbidities (SURMOUNT-MAINTAIN)
Brief Title: A Study of LY3298176 (Tirzepatide) For the Maintenance of Body Weight Reduction in Participants Who Have Obesity or Overweight With Weight-Related Comorbidities
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18720; I8F-MC-GPIQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirzepatide 5 milligram (mg) (Experimental): Participants will receive tirzepatide subcutaneously (SC).
  Interventions: Drug: Tirzepatide
- Tirzepatide Maximum Tolerated Dose (Experimental): Participants will receive tirzepatide SC.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide 5 milligram (mg); Tirzepatide Maximum Tolerated Dose
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of tirzepatide for the maintenance of body weight reduction.

DETAILED DESCRIPTION:
All enrolled participants will complete a 60-week open-label Weight-Loss Period on tirzepatide maximum tolerated dose (MTD) and upon meeting randomization criteria will enter a 52-week double-blinded Weight Maintenance Period to be assigned to either tirzepatide 5 mg, tirzepatide MTD or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) of ≥30 kilogram/square meter (kg/m²) or ≥27 kg/m² and previously diagnosed with at least 1 of the following weight related comorbidities:

  * Hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight (BW)

Exclusion Criteria:

* Have Type 1 Diabetes (T1D) or Type 2 Diabetes (T2D), a history of ketoacidosis, or hyperosmolar state or coma.
* Have a self-reported change in BW>5 kilogram (kg) within 3 months prior to screening
* Have a prior or planned surgical treatment for obesity, excluding liposuction or abdominoplasty if performed >1 year prior to screening.
* Have a history of chronic or acute pancreatitis
* Have any of the following cardiovascular conditions within 3 months prior to week 0.

  * Acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, and hospitalization due to congestive heart failure (CHF)
  * family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Any lifetime history of a suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent Maintenance of Body Weight (BW) Reduction Achieved during the 60-Week Weight Loss Period | Week 112
  Mean percent maintenance of BW reduction achieved during the 60-Week weight loss period will be measured in participants who have reached a BW plateau.

SECONDARY OUTCOMES:
Number of Participants with an Assessment of (yes/no) of Maintaining ≥80% of the BW Reduction Achieved During the 60-week Weight-Loss Period | Week 112
  Assessment of (yes/no) of maintaining ≥80% of the BW reduction achieved during the 60-week weight loss period will be measured in participants who have reached a BW plateau.
Number of Participants with an Assessment of (yes/no) of Maintaining ≥ 15% BW Reduction for Participants Who Have Already Lost ≥15% BW at Randomization | Week 112
  Assessment of (yes/no) of maintaining ≥15% BW reduction for participants who have already lost ≥15% BW at randomization will be measured in participants who have reached a BW plateau.
Percent Change from Baseline in Body Weight | Baseline (Week 0), Week 112
Change from Randomization in Body Weight | Week 60, Week 112
Percent Change from Randomization in Body Weight | Week 60, Week 112
Change from Randomization in Waist Circumference | Week 60, Week 112
Percent Maintenance of BW Reduction Achieved During the 60-week Weight-Loss Period | Week 84

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- United States (20):
  - Cahaba Research - Pelham, Pelham, Alabama
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - New Horizon Research Center, Miami, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Asha Clinical Research - Munster, Hammond, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - L-MARC Research Center, Louisville, Kentucky
  - Prime Health and Wellness/SKYCRNG, Fayette, Mississippi
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Horn DB, Aronne LJ, Wharton S, Bays HE, Gomez-Valderas E, Arad AD, Sharma P, Dunn JP, Senyucel C, Lee CJ. Tirzepatide for the Maintenance of Body Weight Reduction: Rationale, Design, and Baseline Characteristics of SURMOUNT-MAINTAIN. Obesity (Silver Spring). 2025 Oct;33(10):1873-1885. doi: 10.1002/oby.70014. Epub 2025 Sep 7. PMID 40916045
- See also: A Study of LY3298176 (Tirzepatide) For the Maintenance of Body Weight Reduction in Participants Who Have Obesity or Overweight With Weight-Related Comorbidities — https://trials.lilly.com/en-US/trial/424336